CLINICAL TRIAL: NCT00207272
Title: Use of MCT Oil for Enhancement of Weight Loss in Obese Patients-Preliminary Phase 2002-291G
Brief Title: Use of MCT Oil for Enhancement of Weight Loss in Obese Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H-24641
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2008-05-26 (Estimated); Status verified 2008-03

CONDITIONS: Obesity; Weight Loss
Keywords: Hypocaloric MCT oil liquid diet; Hypocaloric LCT oil liquid diet; Visceral and omental adipose tissue; Subcutaneous abdominal adipose tissue; Gastric bypass surgery
MeSH Terms: conditions — Obesity; Weight Loss | interventions — Blood Specimen Collection

INTERVENTIONS:
Behavioral: 1170-1870 kcal/day liquid diet
Procedure: Gastric bypass surgery
Procedure: Biopsy.visceral adipose tissue
Procedure: Biopsy.omental adipose tissue
Procedure: Biopsy. subcutaneous abdominal adipose tissue
Procedure: Blood sample

SUMMARY:
Twelve obese patients approved for gastric bypass surgery will be randomized to either receive an MCT-based or LCT-based liquid diet for a 4 week period. These diets will be identical except for the quality of the fat. The intervention will be double-blinded. Six patients will receive a daily diet consisting of 5 liquid meals using the HMR 800 meal replacement product (Health Management Resources, Inc; 160 calories/shake) with 44.5 grams MCT oil (Life Enhancement Products, Inc., Petaluna, CA; 8.3 kcal/gm) added. Six patients will receive the same HMR diet but with 41 grams LCT oil (corn oil; 9 kcal/gm) added. Patients in both groups will be given a list of supplemental foods that are suitable for the study. They may choose to eat up to an additional 700 kcal per day from this list and will be asked to complete food records for monitoring of their caloric intake. Patients will undergo gastric bypass surgery after 4 weeks of being on their diets. Patients in both groups will be seen weekly by a registered dietitian and a physician. Blood pressure and weight will be recorded, and any adverse events will be noted and cared for as is appropriate. Dietary instruction will be reviewed as needed.Both diets will be 1170-1870 kcal/day, consisting of 36% CHO, 26.2% protein, and 37.6% fat. The MCT diet will contain 30.2% of total calories at MCT oil. The percentages given are based on the shake and oil consumption only (1170 kcal/day). The remainder of the diet will vary according to patients' selections from the list of permitted foods, up to an additional 700 kcal/day (for the total 1870 kcal/day). All subjects will receive a multi-vitamin each day. Subjects will also receive two Fibercon capsules per day to prevent possible bowel changes associated with being on a full liquid diet. During surgery, biopsies of visceral and omental adipose tissue, as well as subcutaneous abdominal adipose tissue, will be obtained. Tissue will be analyzed to determine mRNA levels of key enzymes in fatty acid esterification, lipolysis, and oxidative disposition. This preliminary phase will be conducted to determine whether visceral, omental, and subcutaneous abdominal adipose tissue behave similarly when exposed to an MCT-based diet.

DETAILED DESCRIPTION:
In this the preliminary phase, a total of 12 obese patients who have been accepted to undergo gastric restrictive surgery will be recruited. Although the inclusion criteria for the secondary companion pilot study include diabetic patients, having diabetes mellitus is not necessary for the testing of the hypothesis in the preliminary phase. The aim is to test whether subcutaneous adipose tissue in the abdominal region is similar to visceral and omental adipose tissue in terms of cellular mechanisms after ingestion of MCT oil.

Twelve obese patients approved for gastric bypass surgery will be randomized to either receive an MCT-based or LCT-based liquid diet for a 4 week period. These diets will be identical except for the quality of the fat. The intervention will be double-blinded. Six patients will receive a daily diet consisting of 5 liquid meals using the HMR 800 meal replacement product (Health Management Resources, Inc; 160 calories/shake) with 44.5 grams MCT oil (Life Enhancement Products, Inc., Petaluna, CA; 8.3 kcal/gm) added. Six patients will receive the same HMR diet but with 41 grams LCT oil (corn oil; 9 kcal/gm) added. Patients in both groups will be given a list of supplemental foods that are suitable for the study. They may choose to eat up to an additional 700 kcal per day from this list and will be asked to complete food records for monitoring of their caloric intake. Patients will undergo gastric bypass surgery after 4 weeks of being on their diets. Patients in both groups will be seen weekly by a registered dietitian and a physician. Blood pressure and weight will be recorded, and any adverse events will be noted and cared for as is appropriate. Dietary instruction will be reviewed as needed.

Both diets will be 1170-1870 kcal/day, consisting of 36% CHO, 26.2% protein, and 37.6% fat. The MCT diet will contain 30.2% of total calories at MCT oil. The percentages given are based on the shake and oil consumption only (1170 kcal/day). The remainder of the diet will vary according to patients' selections from the list of permitted foods, up to an additional 700 kcal/day (for the total 1870 kcal/day). Subjects will receive a multi-vitamin each day. Subjects will also receive two Fibercon capsules per day to prevent possible bowel changes associated with being on a full liquid diet. It is estimated patients will lose between 10 and 30 pounds before surgery. This is a standard of care as all patients are encouraged to lose this amount prior to surgery. This small amount of weight loss from initial body weight is considered beneficial in reducing complications of gastric bypass surgery in morbidly obese patients with significant co-morbidities.

During surgery, biopsies of visceral and omental adipose tissue, as well as subcutaneous abdominal adipose tissue, will be obtained. Tissue will be analyzed to determine mRNA levels of key enzymes in fatty acid esterification, lipolysis, and oxidative disposition. This preliminary phase will be conducted to determine whether visceral, omental, and subcutaneous abdominal adipose tissue behave similarly when exposed to an MCT-based dietIn Phase 1 and 2, these results will be used to extrapolate effects on visceral and omental adipose tissue from effects seen on subcutaneous adipose tissue.

In addition, small samples of the tissue (approximately .25 cm x .25cm) for each of the 12 subjects will be shipped to Quantomix, where the samples will be viewed under electron microscopy. There will be no additional tissue removed in the OR for this, and there will be no added risk to the subjects. Quantomix will not receive any identifying information on the samples; therefore there will be no breach of confidentiality.

STUDY PROCEDURES: Screening for Preliminary Phase Twelve obese subjects will be recruited from the Nutrition and Weight Management Center population of gastric restrictive surgery patients. The subjects will have met all requirements for and received prior approval for the gastric restrictive surgery. The patient will sign the IRB-approved Informed Consent - Surgical Intervention form at the Baseline visit. Inclusion criteria includes age 18-65 years and BMI >40 kg/m2 or >35 kg/m2 with co-morbidities. Exclusions are those that are a part of the normal standard of care in the pre-selection process for approval of surgery, clinically severe lactose intolerance, alcohol dependence, and a significant egg allergy.

Baseline and Remaining Visits The Baseline visit will be within two weeks of the screening visit. For the procedures to be performed at the baseline and weekly visits, see Table A attached.

Procedure for subcutaneous adipose tissue needle biopsy The surgeon will remove three pieces of fat tissue measuring 2 inches x 2 inches x 2 inches from the fat under the skin during the gastric restrictive surgery. In the surgical field, it is appropriate to remove this large of a piece of tissue in order to be able to extrapolate and define how much tissue will be required to be removed by punch biopsy in Phase 1 and 2 of the secondary companion study (in the secondary companion study, it is expected that 100 mg subcutaneous tissue will yield 3 micrograms of total RNA. The amount of tissue removed during surgery will be greater than that amount to ensure the projected yield). The surgeon will also remove two pieces of fat tissue from the abdomen during surgery. In total, one piece will be taken from the fat tissue covering the stomach (omental), one piece from just under the skin (subcutaneous), and the other piece from the fat tissue covering the bowels or intestines (visceral). These are fat tissues that are in the area that the surgery will be performed. The biopsy will not interfere in any way with the surgery. The surgeon will also draw a sample of blood (12 mL) to be used for hematology, serum chemistry, hemoglobin A1C, serum lipids, thyroid function test, serum insulin, serum hydroxybutyrate (possibly elevated in MCT-fed subjects), serum leptin, and serum free fatty acid concentration. The surgeon will explain all of this to the subject prior to surgery.

Study schedule:

Pre-Op Diet:

1. Prior to the gastric restrictive surgery, eligible patients will receive dietary instructions by a registered dietitian for a daily diet consisting of 5 liquid meals using the HMR 800 meal replacement product (Health Management Resources, Inc.) with 44.5 grams MCT oil or 41 grams LCT oil added. Patients in both groups will be given a list of supplemental foods that are suitable for the study. They may choose to eat up to an additional 700 kcal per day from this list and will be asked to complete food records for monitoring of their caloric intake. Depending on how much food each patient eats, this will be a daily caloric intake of approximately 1170-1870 calories. All patients will be instructed to refrain from any alcohol intake while in the study.
2. All patients will undergo gastric bypass surgery after 4 weeks of MCT oil/HMR or LCT oil/HMR.

Post-Op Diet:

Following surgery, subjects will follow the usual standard of care implemented in the Nutrition and Weight Management Clinic through post-operative visits with the surgeon and registered dietitian. Diet Stages Following Gastric Restrictive Surgery is attached hereto as Appendix A.

Biopsy Procedure:

1.During gastric restrictive surgery, biopsies of visceral and omental adipose tissue as well as subcutaneous abdominal adipose tissue will be obtained.

The surgeon will remove three pieces of fat tissue measuring 2 inches x 2 inches x 2 inches from the fat under the skin during the gastric restrictive surgery. In the surgical field, it is appropriate to remove this large of a piece of tissue in order to be able to extrapolate and define how much tissue will be required to be removed by punch biopsy in Phase 1 and 2 of the secondary companion study (In the secondary companion study, it is expected that 100 mg subcutaneous tissue will yield 3 micrograms of total RNA. The amount of tissue removed during surgery will be greater than that amount to ensure the projected yield). The surgeon will also remove two pieces of fat tissue from the abdomen during surgery. In total, one piece will be taken from the fat tissue covering the stomach (omental), one piece from just under the skin (subcutaneous), and the other piece from the fat tissue covering the bowels or intestines (visceral). These are fat tissues that are in the area that the surgery will be performed. The biopsy will not interfere in any way with the surgery. The surgeon will also draw a sample of blood to be used for hematology, serum chemistry, hemoglobin A1C, serum lipids, thyroid function test, serum insulin, serum hydroxybutyrate (possibly elevated in MCT-fed subjects), serum leptin, and serum free fatty acid concentration. The surgeon will explain all of this to the subject prior to surgery.

Screening period (up to 2 weeks)

1. Prior to the Screening visit, in the pre-operative visit, the Preliminary Phase will be explained to patients who have been pre-approved for gastric restrictive surgery. Questions will be answered at that time.
2. Initial screening form will be completed
3. Pre-approval for gastric restrictive surgery will be documented.
4. IRB-approved written consent form, signed at the pre-operative visit with the surgeon co-investigator and medical co-investigator will be documented.
5. Patient will be scheduled to return for Baseline visit if eligible for study.

Baseline (within 2 weeks of screening) ± 4 days. Beginning of the study will be within 2-3 weeks after screening visit.

1. Fasting blood samples will be obtained for hematology, serum chemistry, hemoglobin A1C, serum lipids, thyroid function test, serum insulin, serum hydroxybutyrate (possibly elevated in MCT-fed subjects), serum leptin, and serum free fatty acid concentration.
2. Weight and blood pressure will be recorded.
3. Study diet and instructions will be dispensed.
4. Patient will be scheduled for surgery at the end of Week 4 of the study diet.

Weekly visits (with registered dietitian and physician)

1. Weight and blood pressure will be recorded.
2. Dietary instruction will be reviewed as necessary.
3. Adverse effects will be noted.
4. Study diet will be dispensed as needed.
5. At the visit with the dietitian and physician one day before the gastric bypass surgery, blood samples will again be obtained for hematology, serum chemistry, hemoglobin A1C, serum lipids, thyroid function test, serum insulin, serum hydroxybutyrate (possibly elevated in MCT-fed subjects), serum leptin, and serum free fatty acid concentration.

Unscheduled visits (UV):

If necessary for patient safety, unscheduled visits may be arranged. Unscheduled source document sets used for visits attended between routine patient visits will be labeled with the last attended visit number followed by a decimal point and the number of the unscheduled visit (i.e. if two unscheduled visits are attended between Week 0 and Week 1 then those unscheduled visits would be labeled as unscheduled visit sets 0.1 and 0.2 in chronological order).

At unscheduled visits the following shall be completed as indicated:

* Blood samples will be collected for laboratory evaluation, if clinically indicated.
* Adverse events will be documented.
* A physical examination will be performed, if clinically indicated.
* An ECG will be performed, if clinically indicated.

ELIGIBILITY:
Inclusion Criteria:

* Approved for gastric bypass surgery
* Age: 18-65 years
* Gender: Male and female
* BMI: >40 kg/m2 or >35 kg/m2
* Obesity associated co-morbidities
* Race: All

Exclusion Criteria:

* Those that are a part of the normal standard of care in the pre-selection process for approval of surgery
* Clinically severe lactose intolerance
* Alcohol dependence
* Egg allergy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2003-07; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
To determine if the influence that MCFA have on the expression of genes that modulate lipid metabolism in adipose tissue is the same regardless of adipose fat depot

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Apovian, MD, Principal Investigator — Boston University Medical Cneter; Sherman Bigornia, Study Chair — Boston University; James Kirkland, MD,PhD, Study Chair — Boston University; Peter Burke, MD, Study Chair — Boston University; Wen Guo, PhD, Study Chair — Boston University; Robert Forse, MD, Study Chair — Boston University; Diana Cullum-Dugan, RD,LD, Study Chair — Boston University; Donald Hess, Study Chair — Boston University
Locations (1):
- Boston University Medical Center, Boston, Massachusetts, United States

REFERENCES:
- [Background] Baba N, Bracco EF, Hashim SA. Enhanced thermogenesis and diminished deposition of fat in response to overfeeding with diet containing medium chain triglyceride. Am J Clin Nutr. 1982 Apr;35(4):678-82. doi: 10.1093/ajcn/35.4.678. PMID 7072620
- [Background] Guo W, Choi JK, Kirkland JL, Corkey BE, Hamilton JA. Esterification of free fatty acids in adipocytes: a comparison between octanoate and oleate. Biochem J. 2000 Jul 15;349(Pt 2):463-71. doi: 10.1042/0264-6021:3490463. PMID 10880345
- [Background] Geliebter A, Torbay N, Bracco EF, Hashim SA, Van Itallie TB. Overfeeding with medium-chain triglyceride diet results in diminished deposition of fat. Am J Clin Nutr. 1983 Jan;37(1):1-4. doi: 10.1093/ajcn/37.1.1. PMID 6849272
- [Background] Bray GA, Lee M, Bray TL. Weight gain of rats fed medium-chain triglycerides is less than rats fed long-chain triglycerides. Int J Obes. 1980;4(1):27-32. PMID 7390698
- [Background] Han J, Farmer SR, Kirkland JL, Corkey BE, Yoon R, Pirtskhalava T, Ido Y, Guo W. Octanoate attenuates adipogenesis in 3T3-L1 preadipocytes. J Nutr. 2002 May;132(5):904-10. doi: 10.1093/jn/132.5.904. PMID 11983812
- [Background] Krotkiewski M. Value of VLCD supplementation with medium chain triglycerides. Int J Obes Relat Metab Disord. 2001 Sep;25(9):1393-400. doi: 10.1038/sj.ijo.0801682. PMID 11571605
- [Background] Tsuji H, Kasai M, Takeuchi H, Nakamura M, Okazaki M, Kondo K. Dietary medium-chain triacylglycerols suppress accumulation of body fat in a double-blind, controlled trial in healthy men and women. J Nutr. 2001 Nov;131(11):2853-9. doi: 10.1093/jn/131.11.2853. PMID 11694608
- [Background] Bendixen H, Flint A, Raben A, Hoy CE, Mu H, Xu X, Bartels EM, Astrup A. Effect of 3 modified fats and a conventional fat on appetite, energy intake, energy expenditure, and substrate oxidation in healthy men. Am J Clin Nutr. 2002 Jan;75(1):47-56. doi: 10.1093/ajcn/75.1.47. PMID 11756059
- [Background] Papamandjaris AA, White MD, Raeini-Sarjaz M, Jones PJ. Endogenous fat oxidation during medium chain versus long chain triglyceride feeding in healthy women. Int J Obes Relat Metab Disord. 2000 Sep;24(9):1158-66. doi: 10.1038/sj.ijo.0801350. PMID 11033985
- [Background] St-Onge MP, Jones PJ. Physiological effects of medium-chain triglycerides: potential agents in the prevention of obesity. J Nutr. 2002 Mar;132(3):329-32. doi: 10.1093/jn/132.3.329. PMID 11880549